CLINICAL TRIAL: NCT06474728
Title: A Randomised Trial of an Emollient Containing Postbiotic Saccharomyces and Lactobacillus for Improving Clinical Symptoms of Atopic Dermatitis Aged 0-6 Years in Remission
Brief Title: Effects of an Emollient Containing Postbiotic Saccharomyces and Lactobacillus on Pediatric Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADskincare2024
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Atopic Dermatitis; Eczema; Emollient
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Therapeutics; Lacteol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with an Emollient Containing Postbiotic Saccharomyces and Lactobacillus (Experimental)
  Interventions: Other: Treatment with an Emollient Containing Postbiotic Saccharomyces and Lactobacillus
- Treatment without an Emollient Containing Postbiotic Saccharomyces and Lactobacillus (No Intervention)

INTERVENTIONS:
Other: Treatment with an Emollient Containing Postbiotic Saccharomyces and Lactobacillus — Treatment with an Emollient Containing Postbiotic Saccharomyces and Lactobacillus, with the dose of 100g per week,lasting for 12weeks.
  Arms: Treatment with an Emollient Containing Postbiotic Saccharomyces and Lactobacillus

SUMMARY:
The goal of this study is to investigate whether the use of emollients containing postbiotic Saccharomyces and Lactobacillus can significantly reduce the risk of atopic dermatitis (AD) recurrence in pediatric patients aged 0-6 years during the remission phase, compared to the routine maintenance treatment with conventional emollients.

DETAILED DESCRIPTION:
A single-center, randomized, parallel-controlled study was conducted to evaluate the efficacy of an emollient containing postbiotic Saccharomyces and Lactobacillus in 98 children aged 0 to 6 years with moderate AD. Participants were randomly assigned to the experimental group (49 cases) and the control group (49 cases).

During the screening phase, hydrocortisone butyrate cream or desoximetasone cream was topically applied twice daily to the affected areas, along with the emollient twice daily for 2 to 4 weeks until the Investigator's Global Assessment (IGA) score was ≤1, indicating entry into the intervention phase. In the intervention phase, the experimental group discontinued the corticosteroid creams and continued with the emollient twice daily, while the control group discontinued both medication and emollient.

The recurrence of AD, Eczema Area and Severity Index (EASI), Infant/Child Dermatology Quality of Life Index (IDQOL/CDQOL), and adverse events were assessed at weeks 4, 8, and 12 of the intervention phase. Additionally, non-invasive measurements of skin barrier function were conducted, including:

Transepidermal water loss (TEWL) to assess water loss from the skin. Skin electrical capacitance to measure water retention in the stratum corneum. Skin pH to determine the skin's acidity level.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must meet the diagnostic criteria established by Williams.
2. Moderate atopic dermatitis is defined by an Eczema Area and Severity Index (EASI) score of 7.1 to 21.0, and an Investigator's Global Assessment (IGA) score between 2 and 3.
3. Age range is 0 to 6 years, with no gender restrictions.
4. Guardians of the participants must be willing to apply the test product to the participants as directed by the physician throughout the study period.
5. Participants should not have received topical medication within 14 days prior to enrollment, including calcineurin inhibitors (e.g., topical tacrolimus or pimecrolimus), corticosteroid formulations, or topical antihistamines.
6. Within 4 weeks prior to enrollment, participants should not have received non-steroidal immunosuppressants (e.g., cyclosporine, methotrexate) or phototherapy, nor should they have used systemic corticosteroids or systemic antihistamines.
7. Participants are not allowed to use other similar products during the entire study period.
8. Prior to the commencement of any study-specific examination or procedural step, participants must sign an informed consent form. For infants and young children aged 0 to 6 years, the guardians must sign an informed consent waiver on behalf of the child and also sign a parental version of the informed consent form.

Exclusion Criteria:

1. Do not meet the diagnostic criteria established by Williams.
2. Children with acute exacerbation characterized by erosion, exudation, or secondary infection.
3. Presence of open skin infections (bacterial, viral, or fungal) at the application site.
4. Children currently participating in other clinical studies or having participated within the last 3 months.
5. Children who have received topical medication within 14 days prior to enrollment, including calcineurin inhibitors (e.g., topical tacrolimus or pimecrolimus), corticosteroid formulations, or topical antihistamines.
6. Children who have received non-steroidal immunosuppressants (e.g., cyclosporine, methotrexate) or phototherapy, systemic corticosteroids, or systemic antihistamines within 4 weeks prior to enrollment.
7. Children with severe immune system disorders (such as lymphoma, AIDS, Wiskott-Aldrich syndrome) or a history of malignant tumors.
8. Children with severe heart, liver, or kidney diseases.
9. Children with other skin diseases in the treatment area besides atopic dermatitis.
10. Known allergy to hydrocortisone butyrate cream or the test product.
11. Poor compliance of the subject, known inability to attend visits on time, or unwillingness to comply with the study protocol during the study period.
12. Any condition or previous/concurrent treatment that makes the subject ineligible for this study.

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-01-06 (Actual); Study Completion 2026-01-06 (Actual)

PRIMARY OUTCOMES:
Recurrence rate during the intervention phase | 12 weeks
  During the intervention phase, when the patient's Investigator's Gobal Assessment (lGA) score reaches 2 or higher, the investigators defined it as recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology,Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang S, Wang L, Li P, Shu H, Shen C, Wu Y, Luo Z, Miao L, Wang H, Jiao L, Tian J, Peng X, Zhao M, Liu Y, Nie X, He L, Ma L. The improvement of infantile atopic dermatitis during the maintenance period: A multicenter, randomized, parallel controlled clinical study of emollients in Prinsepia utilis Royle. Dermatol Ther. 2020 Mar;33(2):e13153. doi: 10.1111/dth.13153. Epub 2019 Nov 22. PMID 31705602
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31705602/